CLINICAL TRIAL: NCT06034158
Title: Molecular Basis of Loss Aversion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Tang, Deputy Chief Physician, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20230496
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Healthy
MeSH Terms: interventions — benserazide, levodopa drug combination; Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- madopar-propranolol-placebo (Other): In a within-subjects design, participants will take madopar, propranolol, and placebo each once in three separate sessions.
  Interventions: Drug: single-dose madopar, single-dose propranolol, and single-dose placebo by order
- madopar-placebo-propranolol (Other): In a within-subjects design, participants will take madopar, placebo, and propranolol each once in three separate sessions.
  Interventions: Drug: single-dose madopar, single-dose placebo, and single-dose propranolol by order
- propranolol-madopar-placebo (Other): In a within-subjects design, participants will take propranolol, madopar, and placebo each once in three separate sessions.
  Interventions: Drug: single-dose propranolol, single-dose madopar, and single-dose placebo by order
- propranolol-placebo-madopar (Other): In a within-subjects design, participants will take propranolol, placebo, and madopar each once in three separate sessions.
  Interventions: Drug: single-dose propranolol, single-dose placebo, and single-dose madopar by order
- placebo-propranolol-madopar (Other): In a within-subjects design, participants will take placebo, propranolol, and madopar each once in three separate sessions.
  Interventions: Drug: single-dose placebo, single-dose propranolol, and single-dose madopar by order
- placebo-madopar-propranolol (Other): In a within-subjects design, participants will take placebo, madopar, and propranolol each once in three separate sessions.
  Interventions: Drug: single-dose placebo, single-dose madopar, and single-dose propranolol by order

INTERVENTIONS:
Drug: single-dose madopar, single-dose propranolol, and single-dose placebo by order — Participants will take madopar, propranolol, and placebo (orange juice) each once in three separate sessions. The interval between every two sessions will be at least 3 days.
  Arms: madopar-propranolol-placebo
Drug: single-dose madopar, single-dose placebo, and single-dose propranolol by order — Participants will take madopar, placebo(orange juice), and propranolol each once in three separate sessions. The interval between every two sessions will be at least 3 days.
  Arms: madopar-placebo-propranolol
Drug: single-dose propranolol, single-dose madopar, and single-dose placebo by order — Participants will take propranolol, madopar, and placebo(orange juice) each once in three separate sessions. The interval between every two sessions will be at least 3 days.
  Arms: propranolol-madopar-placebo
Drug: single-dose propranolol, single-dose placebo, and single-dose madopar by order — Participants will take propranolol, placebo(orange juice), and madopar each once in three separate sessions. The interval between every two sessions will be at least 3 days.
  Arms: propranolol-placebo-madopar
Drug: single-dose placebo, single-dose propranolol, and single-dose madopar by order — Participants will take placebo(orange juice), propranolol, and madopar each once in three separate sessions. The interval between every two sessions will be at least 3 days.
  Arms: placebo-propranolol-madopar
Drug: single-dose placebo, single-dose madopar, and single-dose propranolol by order — Participants will take placebo(orange juice), madopar, and propranolol each once in three separate sessions. The interval between every two sessions will be at least 3 days.
  Arms: placebo-madopar-propranolol

SUMMARY:
The goal of this clinical trial is to test the roles of dopamine and norepinephrine in decision making related to loss aversion in the healthy population. The main question it aims to answer is whether temporarily boosting dopamine activity or temporarily suppressing norepinephrine activity has an impact on processing of potential gains and losses in financial decision making, social decision making, transaction decision making and moral decision making. Accordingly, participants will complete four decision-making tasks, namely investment task, driving task, trading task, and die task, after taking madopar, propranolol or placebo. Participants' psychological traits and psychiatric symptoms will be assessed once they are enrolled before the first-session day.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-40 years old (including boundary value).
2. Elementary school education or above, able to understand the research content.
3. Body temperature, blood pressure, heart rate, respiratory rate, and electrocardiogram are all normal. Among them, the blood pressure range is 100-139/70-89 mmHg, and the heart rate range is 60-85 beats/min.

Exclusion Criteria:

1. Vulnerable groups, including people with mental illness, cognitive impairment, critically ill subjects, minors, pregnant women, illiterates, etc.
2. Family history of genetic diseases.
3. Major physical diseases, including cardiovascular, respiratory, digestive, renal, endocrine, blood and other systemic diseases.
4. History of alcohol/drug dependence.
5. Lactating women.
6. The cardiopulmonary function test results are poor.
7. Have ever taken madopar or propranolol for medical use.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Choices to invest or not in the investment task | between 1-2 hours after taking the drugs or the placebo
  Participants decide whether or not to accept investment options that entail a 50/50 chance of winning some amount of money and losing some amount of money.
Response times to invest or not in the investment task | between 1-2 hours after taking the drugs or the placebo
  Participants decide whether or not to accept investment options that entail a 50/50 chance of winning some amount of money and losing some amount of money.
Choices to turn or not in the driving task | between 1-2 hours after taking the drugs or the placebo
  Participants decide whether or not to make turns during driving in order to sacrifice some number of person(s) to save some number of person(s) .
Response times to turn or not in the driving task | between 1-2 hours after taking the drugs or the placebo
  Participants decide whether or not to make turns during driving in order to sacrifice some number of person(s) to save some number of person(s) .
Choices to buy or sell in the trading task | between 1-2 hours after taking the drugs or the placebo
  Participants decide whether or not to buy or sell a product at certain prices.
Response times to buy or sell in the trading task | between 1-2 hours after taking the drugs or the placebo
  Participants decide whether or not to buy or sell a product at certain prices.
Reported outcomes in die task | between 1-2 hours after taking the drugs or the placebo
  Participants report the outcome for each throw of the die.

SECONDARY OUTCOMES:
Affects | before and 1 hour after taking the drugs or the placebo
  Participants' affects will be assessed using the Positive and Negative Affective Scale (PANAS).Scores can range from 10 to 50 for both the Positive and Negative Affect, with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheng F, Ramakrishnan A, Seok D, Zhao WJ, Thelaus S, Cen P, Platt ML. Decomposing loss aversion from gaze allocation and pupil dilation. Proc Natl Acad Sci U S A. 2020 May 26;117(21):11356-11363. doi: 10.1073/pnas.1919670117. Epub 2020 May 8. PMID 32385152